CLINICAL TRIAL: NCT00982332
Title: Efficacy of Micro-pulse Steroid Therapy as Induction Therapy in Patients With Polymyalgia Rheumatica
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Gleb Slobodin MD, Bnai Zion MC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: POLYMYALGIA1
Record Dates: First submitted 2009-09-15; First posted 2009-09-23 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Polymyalgia Rheumatica
Keywords: polymyalgia rheumatica
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — Betamethasone; betamethasone dipropionate, betamethasone sodium phosphate drug combination; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- betamethasone (Active Comparator): patients treated with a single intramuscular injection of betamethasone
  Interventions: Drug: Betamethasone; Drug: isotonic sodium chloride solution (placebo)
- isotonic sodium chloride solution (Placebo Comparator)
  Interventions: Drug: isotonic sodium chloride solution (placebo)

INTERVENTIONS:
Drug: Betamethasone — betamethasone dipropionate 20 mg + betamethasone sodium phosphate 8 md as a single intramuscular injection
  Other Names: diprospan injection
  Arms: betamethasone
Drug: isotonic sodium chloride solution (placebo) — 4 ml intramuscular

SUMMARY:
The study will examine the efficacy of a single intramuscular injection of betamethasone dipropionate/betamethasone sodium phosphate at the dose of 20mg/8mg (injection volume 4 ml) as an induction therapy in patients with polymyalgia rheumatica. Twenty patients will be randomized to receive an injection of betamethasone or placebo (isotonic NaCl solution) immediately after diagnosis. Both groups will receive the standard-of-care steroid therapy, starting from 10 mg of prednisone every day (qd), tapered down by 2.5 mg monthly if the disease is not active (scheduled monthly follow-ups by a rheumatologist). Primary outcome measures: the total cumulative dose of glucocorticosteroids and disease duration.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of polymyalgia rheumatica

Exclusion Criteria:

* decompensated diabetes mellitus
* decompensated arterial hypertension

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-09 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
a total dose of glucocorticoids used in the course of the disease | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel